CLINICAL TRIAL: NCT02055352
Title: 24-week Study to Evaluate Efficacy and Safety of the Combination Budesonide / Indacaterol vs Fluticasone / Salmeterol in Patients With COPD
Brief Title: Study to Evaluate Efficacy/Safety of Combination Budesonide/Indacaterol vs Fluticasone/Salmeterol in Patients With COPD
Acronym: COMBINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQAB149BAR01
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Fluticasone; indacaterol; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide/indacaterol (Experimental): Participants will receive a fixed combination of fluticasone and salmeterol during 4 weeks followed by a free combination of budesonide and indacaterol for the remainig of study.
  Interventions: Drug: Budesonide; Drug: Fluticasone; Drug: Indacaterol; Drug: Salmeterol
- Fluticasone / salmeterol (Active Comparator): Fixed combination of fluticasone and salmeterol
  Interventions: Drug: Fluticasone; Drug: Salmeterol

INTERVENTIONS:
Drug: Budesonide — Budesonide 400 mcg twice a day via Breezhaler® device
  Arms: Budesonide/indacaterol
Drug: Fluticasone — Fluticasone 250 mcg twice daily via Accuhaler® device
Drug: Indacaterol — Indacaterol 150 mcg once daily via Breezhaler® device
  Arms: Budesonide/indacaterol
Drug: Salmeterol — Salmeterol 50 mcg twice daily via Diskus® device

SUMMARY:
To demonstrate the free combination of budesonide and indacaterol is as efficacious as fluticasone and salmeterol in patients with COPD

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed
* Outpatients with stable COPD groups C and D according to the 2011 GOLD Guidelines.
* Current or ex-smokers who have a smoking history of at least 10 pack years
* Patients with a history of at least one exacerbation.
* Patients able to read and complete

Exclusion Criteria:

* Use of other investigational drugs within 30 days
* Patients with a history of hypersensitivity to any of the study drugs
* History or current diagnosis of ECG abnormalities
* Patients with diabetes Type I or uncontrolled diabetes Type II including patients with a history of blood glucose levels consistently outside the normal range
* Patients who have not achieved an acceptable spirometry result at Visit 1
* Patients with a body mass index (BMI) of more than 40 kg/m2
* Patients with lung cancer or a history of lung cancer
* Patients with a history of malignancy of any organ system
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment
* Patients who do not maintain regular day/night, waking/sleeping cycles (e.g., night shift workers)
* Patients that are uncontrolled or unstable on permitted therapy, who in the opinion of the investigator, have clinically significant renal, cardiovascular, neurological, endocrine, immunological, psychiatric, gastrointestinal, hepatic, or haematological abnormalities which could interfere with the assessment of the efficacy and safety of the study treatment
* Patients requiring oxygen therapy for chronic hypoxemia
* Patients who have had a respiratory tract infection within 6 weeks prior to Visit 1
* Patients with concomitant pulmonary disease, e.g. pulmonary tuberculosis, bronchiectasis, sarcoidosis, interstitial lung disorder or pulmonary hypertension
* Patients with a known diagnosis of Alpha-1 Antitrypsin deficiency.
* Patients with history of lung surgery
* Patients who are participating in the active phase of a supervised pulmonary rehabilitation program.
* Patients with a history of asthma Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2014-05-30 (Actual); Primary Completion 2016-01-26 (Actual); Study Completion 2016-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- Argentina (9):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Florida, Buenos Aires
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Vicente López, Buenos Aires
  - Novartis Investigative Site, Zárate, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Ciudad Autonoma de Bs As
  - Novartis Investigative Site, Santa Rosa, La Pampa Province
  - Novartis Investigative Site, Salta, Salta Province
- Brazil (4):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Bernardo do Campo, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Chile (2):
  - Novartis Investigative Site, Rancagua, Rancagua
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
- Novartis Investigative Site, Santo Domingo, Republica Dominicana, Dominican Republic
- Novartis Investigative Site, Guayaquil, Guayas, Ecuador
- Honduras (2):
  - Novartis Investigative Site, San Pedro Sula, Honduras
  - Novartis Investigative Site, Tegucigalpa, Honduras
- Mexico (2):
  - Novartis Investigative Site, León, Guanajuato
  - Novartis Investigative Site, Mexico City, Mexico City
- Novartis Investigative Site, Panama City, Provincia de Panamá, Panama

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Budesonide/Indacaterol | Fluticasone / Salmeterol
Started | 109 | 113
Per-Protocol Set (PPS) | 108 | 111
Completed | 103 | 96
Not Completed | 6 | 17
Not completed — Adverse Event | 0 | 1
Not completed — Non-eligible | 0 | 1
Not completed — Poor compliance | 1 | 1
Not completed — Death | 1 | 2
Not completed — Patient decision | 1 | 1
Not completed — Use of prohibited treatment | 0 | 3
Not completed — AE, study drug would be detrimental | 1 | 3
Not completed — Withdrawal of informed consent | 1 | 0
Not completed — Reason unknown | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Budesonide/Indacaterol | Fluticasone / Salmeterol | Total
Number analyzed (Participants) | 109 | 113 | 222
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.1 (9) | 67.3 (8.45) | 67.2 (8.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 54 | 95
  Male | 68 | 59 | 127

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (Non-inferiority Analysis).
Description: Forced Expiratory Volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Time Frame: Baseline and week 12
Population: Per-protocol set (PPS) included all patients in the FAS without any major protocol deviations. Major protocol deviations were defined in the validation analysis plan prior to database lock and the unblinding of the study. Patients were analyzed according to the treatment they are randomized to
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Budesonide/Indacaterol | Fluticasone / Salmeterol
Number analyzed (Participants) | 108 | 111
Liters | 0.080 (0.027) | 0.019 (0.028)
Statistical Analysis 1: Comparison: Budesonide/Indacaterol vs Fluticasone / Salmeterol; Test type: Non-Inferiority or Equivalence — A change of 5-10% from baseline values is considered to be clinically important. The estimated adjusted treatment difference for budesonide 400 μg twice a day/ indacaterol 150 μg once daily minus fixed combination of fluticasone/ salmeterol 250/ 50 μg twice daily was displayed along with the associated one-sided 97.5% confidence interval. If the lower limit of this confidence interval was to the right (i.e. above) - 10 mL, then non-inferiority could be claimed; p = 0.004, Mixed effects General linear model

2. Secondary Outcome: Change in Health Status - mMRC
Description: Modified Medical Research Council scale (mMRC) questionnaire will be completed by participants. 0 Not troubled with breathlessness except with strenuous exercise; 1 Troubled by shortness of breath when hurrying on the level or walking up a slight hill; 2 Walks slower than people of the same age on the level because of breathlessness or has to stop for breath when walking at own pace on the level; 3 Stops for breath after walking about 100 yards or after a few minutes on the level; 4 Too breathless to leave the house or breathless when dressing or undressing
Time Frame: Baseline, week 12 and week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Budesonide/Indacaterol | Fluticasone / Salmeterol
Number analyzed (Participants) | 108 | 111
Score on a scale
  Week 12 | 1.452 (0.111) | 1.623 (0.113)
  Week 24 | 1.315 (0.112) | 1.414 (0.115)

3. Secondary Outcome: Change From Baseline in Mean Daily Number of Puffs of Rescue Medication Used Over the 24 Week Treatment
Description: A day with no rescue medication use is defined from the diary data as any day where the patient recorded no rescue medicine use during the previous 12 hours.
Time Frame: 24 weeks
Population: Per-protocol set (PPS) included all patients in the FAS without any major protocol deviations. Major protocol deviations were defined in the validation analysis plan prior to database lock and the unblinding of the study. Patients that were not discontinued before Visit 3 (day 28±3).
Measure: Mean (Standard Deviation); unit: Puffs
Arm/Group | Budesonide/Indacaterol | Fluticasone / Salmeterol
Number analyzed (Participants) | 105 | 105
Puffs | 10.5 (9.53) | 12.9 (12.34)

4. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second at Week 24 (Analysis of Superiority)
Description: Forced Expiratory Volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing.
Time Frame: Baseline and week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Budesonide/Indacaterol | Fluticasone / Salmeterol
Number analyzed (Participants) | 108 | 111
Liters | 0.063 (0.033) | 0.020 (0.034)

5. Secondary Outcome: Change in Health Status - SGRQ-C
Description: St George's Respiratory Questionnaire short version questionnaire will be completed by participants. The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life)
Time Frame: Baseline, week 12 and week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Budesonide/Indacaterol | Fluticasone / Salmeterol
Number analyzed (Participants) | 108 | 111
Score on a scale
  Week 12 | -8.703 (2.006) | -2.334 (2.053)
  Week 24 | -7.787 (2.308) | -2.523 (2.384)

ADVERSE EVENTS:
Groups:
- Budesonide / Indacaterol (A): Budesonide / Indacaterol (A)
- Fluticasone / Salmeterol (B): Fluticasone / Salmeterol (B)
Arm/Group | Budesonide / Indacaterol (A) | Fluticasone / Salmeterol (B)
Serious Adverse Events (participants affected / at risk) | 10/109 | 9/113
Other Adverse Events (participants affected / at risk) | 24/109 | 39/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide / Indacaterol (A) (N=109) | Fluticasone / Salmeterol (B) (N=113)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cor pulmonale (Cardiac disorders) | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Vascular insufficiency (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Budesonide / Indacaterol (A) (N=109) | Fluticasone / Salmeterol (B) (N=113)
Influenza (Infections and infestations) | 6 | 10
Nasopharyngitis (Infections and infestations) | 11 | 10
Urinary tract infection (Infections and infestations) | 3 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6
Headache (Nervous system disorders) | 1 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.